CLINICAL TRIAL: NCT01936064
Title: A Prospective Phase II Randomized, Blinded Study to Demonstrate the Effectiveness of Jobelyn for the Treatment of Breast Cancer Patients.
Brief Title: The Safety and Efficacy of Jobelyn in the Treatment of Breast Cancer Patients
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lagos State University (Other)
Responsible Party: Principal Investigator, Abiodun Popoola, CONSULTANT IN THE DEPARTMENT OF ONCOLOGY LASUTH, Lagos State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LASUTH/09/2012; HEALTH FOREVER PRODUCT LTD (Other Grant/Funding Number: LAGOS STATE UNIVERSITY)
Record Dates: First submitted 2013-05-18; First posted 2013-09-05 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Haematological Abnormality
Keywords: Breast Cancer; Jobelyn; Sorghum bicolor
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Jobelyn + Cyclophosphamide-Epirubicin6 (Active Comparator): Cyclophosphamide- Epirubicin 6 course regimen to be used with Jobelyn
  Interventions: Dietary Supplement: Jobelyn + Cyclophosphamide-Epirubicin6
- Placebo + Cyclophosphamide- Epirubicin 6 (Active Comparator): Routine drugs for treatment of Breast Cancer used with Placebo
  Interventions: Drug: Placebo + Cyclophosphamide - Epirubicin 6

INTERVENTIONS:
Dietary Supplement: Jobelyn + Cyclophosphamide-Epirubicin6 — Jobelyn (dietary Supplement) to be used with Cyclophosphamide-Epirubicin6
  Other Names: Sorghum bicolor extract
  Arms: Jobelyn + Cyclophosphamide-Epirubicin6
Drug: Placebo + Cyclophosphamide - Epirubicin 6 — Routine drugs for the treatment of breast cancer to be used with Placebo
  Other Names: Breast Cancer drugs
  Arms: Placebo + Cyclophosphamide- Epirubicin 6

SUMMARY:
To determine the effective functionality/potency of Jobelyn as an immunologic and haematologic booster in Breast cancer patients (start-off), thus improving the outlook and the quality of life of such patients generally

DETAILED DESCRIPTION:
Breast cancer is one of the most frequent malignant tumor of women in Nigeria. In Nigeria, among the urban women, the numbers of breast cancer patients were increasing annually, both to aging of the population and increase in age-specific incidences. Case control studies in parts of the country have identified the factors such as null parity, late age at marriage, and late age at first pregnancy are important risk factors. It has also been suggested that western dietary influences changed the lifestyle of urban women could be one of the major causes of the slowly rising incidence of breast cancer in Nigeria. Therefore early detection and search for potential anti-tumour compounds are important in the control of breast cancer.Standard treatment modalities have improved the overall outlook and quality of life for women with breast cancer; however, the fact that more than 50% still succumb to disease highlights the need for new therapeutic approaches and identification of new therapeutic targets.

Jobelyn is made from Sorghum bicolor which grows abundantly in many parts of the world. Major component analysis of the raw materials and the finished product showed that the herbal product contains oligomeric and polymeric proanthocyanidin (OPCs) which are a class of flavonoid complexes. They are also referred to as condensed tannins. They were first discovered in 1948 by Jacques Masquelier, who developed and later patented techniques for the extraction of proanthocyanidin from pine needles and grape seeds. They can also be found in apples, coconut, cocoa beans, black currant, green tea, black tea. Cocoa beans contain the highest concentrations.

In preliminary research, proanthocyanidin was reported to have anti-mutagenic activity. Studies also show that proanthocyanidin antioxidant capabilities are 20 times more powerful than vitamin C and 50 times more potent than vitamin E2. They also work directly to help strengthen all the blood vessels and improve the delivery of oxygen to the cells. Having affinity for cell membranes, they provide nutritional support to reduce capillary permeability and fragility. These they owe to their role in stabilization of collagen and maintenance of elastin.

Oligomeric proanthocyanidin helps in cancer treatment by inhibiting the initiation and progress of cancer cells. This is why according to a study, it was found that Jobelyn water extract had a stronger effect on increasing Cluster of Differentiation 69 expression in Natural Killer cells (higher cytotoxic activity) while Jobelyn Ethyl Alcohol extract had the greatest effect on increasing Cluster of Differentiation 69 expression in Natural Killer T-cells, T-cells and monocytes (activation & proliferation). In addition to its selective cytotoxicity property, oligomeric proanthocyanidin may up-regulate certain apoptosis promoter genes and down-regulate apoptosis-inhibitor genes in cancerous cells.

3-Deoxyanthocyanidins are a rare type of flavonoids restricted to a few plant species. They are the major pigments in flowers of sinningia (Sinningia cardinalis) and are found in silk tissues of certain maize lines. Sorghum is the only dietary source for 3-deoxyanthocyanidins, which are present in large quantities in the bran of some cultivars . Many plants use secondary metabolites to protect themselves against pathogen attack. In sorghum, this defense response is an active process resulting in the accumulation of high levels of 3-deoxyanthocyanidin phytoalexins in infected tissues. Luteolinidin and apigeninidin are the two major 3-deoxyanthocyanidins. Flavonoids are increasingly recognized for their range of health benefits, such as reducing the risks of cardiovascular diseases and cancers due to their antioxidant, anti-inflammatory, and chemoprotective properties. In particular, anthocyanins and anthocyanidins from different sources were shown to suppress proliferation and induce apoptosis in cancer cell lines. In a recent study, 3-deoxyanthocyanidins were found to have antioxidant properties similar to those of anthocyanins, but they are more stable to power of hydrogen, temperature, and light changes,suggesting that they could serve as an alternative source of natural pigments with nutraceutical properties.

The unique properties of 3-deoxyanthocyanidins may extend to their biochemical activity as well. For example, Shih et al. recently demonstrated that the major sorghum 3-deoxyanthocyanidins aglycons, apigeninidin and luteolinidin, were more cytotoxic to human cancer cells than their anthocyanidin analogues, cyanidin and pelargonidin

Recent research publication confirmed that the variety of Sorghum bicolor from which Jobelyn was produced contained two unique compounds which are being reported for the first time in Sorghum and in nature and these compounds have been tested in vitro for their anti-inflammatory properties using Ibuprofen as control. They showed superior results to Ibuprofen for their safety and efficacy properties. Hitherto, 3-deoxyanthocyanidins which have been known to contain two main compounds, apigeninidin and luteolinidin has now been increased to four compounds, courtesy of the two new additions discovered from the unique Sorghum variety which is the main ingredient of Jobelyn.

Anaemia, commonly defined as a haemoglobin level of <14g/dl in men and <12g/dl in women, occurs in over 30% of cancer patients at any point in time, and its incidence increases with treatment and disease progression. This anaemia could be related to the patient (haemoglobinopathies, gastrointestinal problems, thalassemia, etc.), related to the disease (bone marrow infiltration, bowel resection, hypersplenism, diminished nutritional state) or related to therapy (drug-induced haemolysis, hypoplasia of bone marrow-bearing areas such as the pelvis secondary to radiotherapy, bone marrow and renal toxicity secondary to chemotherapy, etc.). Inflammatory cytokines such as tumour necrotic factor-alpha and interleukin-6, among others, play a major role in the pathophysiology of anaemia in the cancer patient, not only through complex mechanisms of the purely inflammatory situation but also through genetic regulatory aspects of erythropoiesis.

Oxidative stress brought about by overwhelming of the body by free radicals from the disease itself (cancer) and the therapy both contribute to increased haemolysis and immune depression, as these degrade cell linings and disrupt many biochemical pathways. Jobelyn, which contains majorly oligomeric proanthocyanidin, prevent cell membrane damage by disrupting the biochemical formation of free radicals, thus preventing the release of haemolytic inflammatory cytokines.

In tandem, by mopping up free radicals, it would be found useful in delaying the onset of opportunistic infection in cancer patients, which in itself can provoke further haemolysis. However, these functions are still being proven in Human Clinical Trials which has so far been carried out in two research centres in Nigeria, though primarily amongst sickle cell and HIV/AIDS patients1. However, this experimental trial is now being extended to cancer patients to assess its usefulness in this condition.

ELIGIBILITY:
Inclusion Criteria:

Women with histologically confirmed breast cancer who had undergone complete or segmental mastectomy plus axillary node dissection were included

Exclusion Criteria:

Patients were excluded if they had distant metastases residual disease in the breast or axilla other serious medical illnesses, or a previous cancer. Women considering pregnancy or using hormones were excluded

Patients who refuse to sign consent form

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-10 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Natural Killer Cells Expression | 6 months
  Evaluation of the expression of activated natural killer cells CD3-CD56+CD69+ after treatment with Jobelyn

SECONDARY OUTCOMES:
Use of health related quality of life measures tool Safety Fractor-36 and self reporting questionnaires | 6 months
  Subjects would use form Safety Fractor-36 to score aspects of well-being
Hematocrit Changes | 6 months
  Changes in levels of hematocrit after treatment with Jobelyn

CONTACTS AND LOCATIONS:
Overall Officials: Abiodun Popoola, M.D., Principal Investigator — Lagos State University
Locations (2):
- Nigeria (2):
  - Lagos State University Teaching Hospital, Ikeja, Lagos
  - Lagos State University, Ikeja, Lagos

REFERENCES:
- [Background] Geera B, Ojwang LO, Awika JM. New highly stable dimeric 3-deoxyanthocyanidin pigments from sorghum bicolor leaf sheath. J Food Sci. 2012 May;77(5):C566-72. doi: 10.1111/j.1750-3841.2012.02668.x. Epub 2012 Apr 10. PMID 22489620
- [Background] Brohan M, Jerkovic V, Collin S. Potentiality of red sorghum for producing stilbenoid-enriched beers with high antioxidant activity. J Agric Food Chem. 2011 Apr 27;59(8):4088-94. doi: 10.1021/jf1047755. Epub 2011 Mar 7. PMID 21381750
- [Background] Yang L, Browning JD, Awika JM. Sorghum 3-deoxyanthocyanins possess strong phase II enzyme inducer activity and cancer cell growth inhibition properties. J Agric Food Chem. 2009 Mar 11;57(5):1797-804. doi: 10.1021/jf8035066. PMID 19256554
- [Background] Kayode AP, Nout MJ, Linnemann AR, Hounhouigan JD, Berghofer E, Siebenhandl-Ehn S. Uncommonly high levels of 3-deoxyanthocyanidins and antioxidant capacity in the leaf sheaths of dye sorghum. J Agric Food Chem. 2011 Feb 23;59(4):1178-84. doi: 10.1021/jf103963t. Epub 2011 Jan 25. PMID 21322653
- [Background] Shih CH, Siu SO, Ng R, Wong E, Chiu LC, Chu IK, Lo C. Quantitative analysis of anticancer 3-deoxyanthocyanidins in infected sorghum seedlings. J Agric Food Chem. 2007 Jan 24;55(2):254-9. doi: 10.1021/jf062516t. PMID 17227050
- [Background] Camargo Filho I, Cortez DA, Ueda-Nakamura T, Nakamura CV, Dias Filho BP. Antiviral activity and mode of action of a peptide isolated from Sorghum bicolor. Phytomedicine. 2008 Mar;15(3):202-8. doi: 10.1016/j.phymed.2007.07.059. Epub 2007 Sep 24. PMID 17890069
- [Background] Burdette A, Garner PL, Mayer EP, Hargrove JL, Hartle DK, Greenspan P. Anti-inflammatory activity of select sorghum (Sorghum bicolor) brans. J Med Food. 2010 Aug;13(4):879-87. doi: 10.1089/jmf.2009.0147. PMID 20673059
- [Background] Park JH, Darvin P, Lim EJ, Joung YH, Hong DY, Park EU, Park SH, Choi SK, Moon ES, Cho BW, Park KD, Lee HK, Kim MJ, Park DS, Chung IM, Yang YM. Hwanggeumchal sorghum induces cell cycle arrest, and suppresses tumor growth and metastasis through Jak2/STAT pathways in breast cancer xenografts. PLoS One. 2012;7(7):e40531. doi: 10.1371/journal.pone.0040531. Epub 2012 Jul 6. PMID 22792362
- [Background] Wu L, Huang Z, Qin P, Yao Y, Meng X, Zou J, Zhu K, Ren G. Chemical characterization of a procyanidin-rich extract from sorghum bran and its effect on oxidative stress and tumor inhibition in vivo. J Agric Food Chem. 2011 Aug 24;59(16):8609-15. doi: 10.1021/jf2015528. Epub 2011 Jul 29. PMID 21780844
- [Background] Devi PS, Kumar MS, Das SM. Evaluation of antiproliferative activity of red sorghum bran anthocyanin on a human breast cancer cell line (mcf-7). Int J Breast Cancer. 2011;2011:891481. doi: 10.4061/2011/891481. Epub 2011 Oct 16. PMID 22312562
- [Background] Awika JM, McDonough CM, Rooney LW. Decorticating sorghum to concentrate healthy phytochemicals. J Agric Food Chem. 2005 Aug 10;53(16):6230-4. doi: 10.1021/jf0510384. PMID 16076098
- [Background] Benson KF, Beaman JL, Ou B, Okubena A, Okubena O, Jensen GS. West African Sorghum bicolor leaf sheaths have anti-inflammatory and immune-modulating properties in vitro. J Med Food. 2013 Mar;16(3):230-8. doi: 10.1089/jmf.2012.0214. Epub 2013 Jan 5. PMID 23289787
- [Background] Tayo AO, Dosunmu AO, Akinola IO, Adewunmi A, Oloyede OA, Akinbami AA, Osikomaiya BI, Makanjuola SB. An open-label, randomized, parallel-group comparative study of the efficacy of sorghum bicolor extract in preoperative anemia. Nutrition. 2017 Jan;33:113-117. doi: 10.1016/j.nut.2016.05.005. Epub 2016 May 18. PMID 27461168
- [Background] Newly isolated compounds from West African Sorghum bicolor leaf sheaths Jobelyn® show potential in cancer immunosurveillance DOI: http://dx.doi.org/10.14312/2052-4994.2016-6